CLINICAL TRIAL: NCT00424905
Title: Evaluation of the Effects of Enterogermina, 2 Billion Bacillus Clausii Spores, on the Intestinal Flora of Children Antibiotic Treated for Bacterial Upper Respiratory Tract Infections: Open, Pilot Study.
Brief Title: DIAMANTE - Diseases Infectious Analysis Microflora Antibiotic Effect
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Medical Director, Sanofi-aventis administrative office
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PM_L_0199; EudraCT # : 2006-002482-39
Record Dates: First submitted 2007-01-19; First posted 2007-01-22 (Estimated); Last update posted 2008-12-01 (Estimated); Status verified 2008-11

CONDITIONS: Gastrointestinal Diseases
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — clausin peptide, Bacillus clausii

ARMS (2):
- 1 (Experimental): Enterogermina® vials containing 2×109 spores of polyantibiotic resistant Bacillus clausii (test drug)
  Interventions: Drug: Bacillus clausii
- 2 (No Intervention): No treatment (reference group)

INTERVENTIONS:
Drug: Bacillus clausii — 2 Enterogermina vials/day for 12 to 17 days (i.e. during the 5 to 10-days antibiotic treatment and for 7 days thereafter.
  Arms: 1

SUMMARY:
To assess the effects of Bacillus clausii (Enterogermina®) on fecal microbial flora (using Polymerase Chain Reaction - Denaturing Gradient Gel Electrophoresis - PCR-DGGE - Method) in antibiotic-treated children with complicated acute otitis media or beta-hemolytic streptococcal pharyngo-tonsillitis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with persistency of symptoms and requiring antibiotics for bacterial upper respiratory tract infections, i.e. complicated acute otitis media (diagnosed by otoscopic examination) or beta-haemolytic streptococcal pharyngo-tonsillitis (diagnosed by pharyngeal swab and rapid antigen detection test or positive culture);
* Outpatients or patients attending an emergency room for both diagnoses, and inpatients in case of complicated acute otitis media;
* Written informed consent from both parents.

Exclusion Criteria:

* History of clinically significant chronic diseases, or chronic diseases necessitating the use of continuous drug therapies, or of any disease that may interfere with the successful completion or the objectives of the trial;
* Clinical evidence of relevant cardiovascular, respiratory, renal, hepatic, gastrointestinal, hematological, neurological or of any disease that may interfere with the successful completion or the objectives of the trial;
* Use of antibiotics, prebiotics or probiotics (medications or dietetic supplements) in the last 2 weeks prior to study entry;
* Hypersensitivity to the investigational product;
* Subjects enrolled in another trial in the previous three months.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2006-12; Primary Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Changes of microbial composition of fecal bacterial flora by PCR-DGGE analysis. | between samples obtained at baseline and follow-up

SECONDARY OUTCOMES:
Changes from baseline of body weight | During the total study period
Assessment of abdominal symptoms | Daily
Presence of Bacillus clausii spores in feces | after heat shock treatment on selective medium.
Number and rate of patients with GI symptoms and time to first development of symptoms. | recorded in a daily diary card for the total study period

CONTACTS AND LOCATIONS:
Overall Officials: Georges Paizis, MD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Milan, Italy